CLINICAL TRIAL: NCT06985407
Title: Acute and Chronic Effects of Grape Extract on Cardiovascular Response Following Exercise
Brief Title: Grape Extract and Exercise Effects on Blood Pressure
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Castilla-La Mancha (Other)
Collaborators: Alvinesa Natural Ingredients (Unknown)
Responsible Party: Principal Investigator, Felix Morales Palomo, PhD; Principal Investigator, University of Castilla-La Mancha
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: POLYPHENOL-EXER-CARDIOVACULAR
Record Dates: First submitted 2025-05-06; First posted 2025-05-22 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Exercise Response; Blood Pressure Monitoring, Ambulatory; Polyphenol
Keywords: Grape extract; Exercise; Vascular function; Blood Pressure; Polyphenol
MeSH Terms: conditions — Motor Activity | interventions — whole grape extract; Population Groups

STUDY DESIGN:
Intervention Model Description: This study will be a crossover randomized control trial. Twelve sedentary adults (mix of males and females) with elevated blood pressure (i.e., prehypertension) will be recruited and, following preliminary and baseline testing, will perform two conditions in random order: a) control (placebo) and b) grape extract (VinteraTM Premium Red Grape). The randomization will be counterbalanced and stratified by sex, and the design will follow a double-blind design. Then, six participants (3 males and 3 females) will start the control condition, and the other group (3 males and 3 females) will initiate the grape extract condition. Each condition will last 7 days for assessing both acute and chronic effects, and there will be a wash-out period of 7 days.
Who Masked: Participant
Masking Description: Several strategies will be used to ensure the double-blind design. First, both formulations will contain identical inert excipients (such as microcrystalline cellulose, magnesium salts of fatty acids, or silicon dioxide) to ensure indistinguishable taste, smell, and texture. Furthermore, the capsules will be identical in color, size, and shape, using standard materials that prevent distinction of the contents. Both formulations will be non-calorie flavoured, avoiding taste differences, especially if the capsules are accidentally chewed. Furthermore, encapsulation will be performed by a specialized laboratory, such as Alvinesa Natural Ingredients, ensuring a consistent preparation. Finally, the capsules will be distributed in identical packaging without distinctive markings that could compromise the double-blind design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Grape extract (VinteraTM Premium Red Grape) (Experimental)
  Interventions: Dietary Supplement: Grape extract (VinteraTM Premium Red Grape)
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Control (placebo) group

INTERVENTIONS:
Dietary Supplement: Grape extract (VinteraTM Premium Red Grape) — Each condition will last 7 days for assessing both acute and chronic effects, and there will be a wash-out period of 7 days.
  Arms: Grape extract (VinteraTM Premium Red Grape)
Dietary Supplement: Control (placebo) group — Each condition will last 7 days for assessing both acute and chronic effects, and there will be a wash-out period of 7 days.
  Arms: Placebo

SUMMARY:
Exercise and grape extract intake (i.e., polyphenol-rich product) can independently improve blood pressure and endothelial function in prehypertensive individuals. Nevertheless, their combined effects remain unexplored. Furthermore, since the biological pathways targeted by both interventions are similar, they could overlap and be amplified by one another, promoting additive or synergistic effects. Animal model studies have reported that a grape seed extract intake prevents exercise-induced oxidative stress, which could improve vascular dysfunction. Furthermore, as previously reported, a single dose of grape seed extract reduces blood pressure, peripheral vasoconstriction, and heart stress, enhancing O2 delivery during exercise in prehypertensive males. These effects may be partly due to endothelium-dependent vasodilation enhancement. Therefore, it is necessary to understand the potential impact of exercise and grape extract on blood pressure and vascular function in prehypertensive individuals.

ELIGIBILITY:
Inclusion Criteria:

* Sedentary individuals (<120 min·wk-1 of moderate-intensity activity assessed by 7-d IPAQ).
* Aged 25-65 years and BMI 18-35 kg/m2.
* Elevated BP (i.e., prehypertensive; systolic and diastolic BP between 120-139 and/or 80-89 mmHg, respectively)

Exclusion Criteria:

* Weight instability (>5kg change in body mass over last 6 months)
* Pregnant or lactating
* Changes in physical activity over the last 3 months and planning on physical activity, or diet throughout the intervention.
* Untreated cardiovascular or renal disease, peripheral vascular disease, hypertension (≥140 mmHg systolic, or ≥90 mmHg diastolic BP), and any disease associated with exercise intolerance.
* Under pharmacological treatment for any cardiometabolic disease (i.e., hypertension, dyslipidemia or hyperglycemia)
* Currently taking dietary supplements that influence the cardiovascular response (e.g., polyphenols, omega-3 fatty acids, Magnesium, nitrates, L-arginine, red ginseng, natto, ginkgo, CoQ10) or used in the last month.
* Current or recent use (within the past 6 months) of tobacco or nicotine-containing products, or illicit drugs.
* Any medical condition or medication that could introduce bias into the study (e.g. neurological disorders)

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Postexercise systolic and diastolic blood pressure (mmHg) | Acute/chronic effects (0 and 7 days)
  Blood pressure will be measured in triplicated each 5 min during 40 minutes of supine rest.
24-hour ambulatory blood pressure following exercise (mmHg) | Acute/chronic effects (0 and 7 days)
  Ambulatory blood pressure will be assessed for 24 hours.
Brachial flow-mediated dilation (%) | Acute/chronic effects (0 and 7 days)
  Flow-mediated dilation (FMD) in the brachial artery will be performed via two-dimensional (2-D)/Doppler ultrasound.
Brachial blood flow (ml·min-1) | Acute/chronic effects (0 and 7 days)
  Brachial artery blood flow will be assessed via 2-D/Doppler ultrasound. Each blood flow recording period will be at least 4 min long.

SECONDARY OUTCOMES:
Postexercise heart rate (bpm) | Acute/chronic effects (0 and 7 days)
  Post-exercise heart rate will be assessed for 40 minutes after completing the exercise.
Plasma nitric oxide concentrations (μmol L-1) | Acute/chronic effects (0 and 7 days)
  Plasma nitric oxide concentrations will be determined using the enzymatic conversion of nitrate to nitrite by nitrate reductase (Thermoscientific; intra-and interassay CV 1.4%- 3.5%).
Circulating endothelial biomarkers | Acute/chronic effects (0 and 7 days)
  Serum E-selectin concentration (ng mL-1); Serum P-selection concentration (ng mL-1); Serum Intracellular adhesion molecule 1 (ICAM-1) concentration (ng mL-1); Serum Vascular cell adhesion molecule 1 (VCAM-1) concentration (ng mL-1); Serum Tissue plasminogen activator (tPA) concentration (ng mL-1)
Exercise total carbohydrate oxidation (g min-1) | Acute/chronic effects (0 and 7 days)
  Total whole-body carbohydrate rates were calculated using non-protein Péronnet and Massicotte's equations
Exercise total fat oxidation (g min-1) | Acute/chronic effects (0 and 7 days)
  Total whole-body fat oxidation rates were calculated using non-protein Péronnet and Massicotte's equations
Heart rate during exercise (bpm) | Acute/chronic effects (0 and 7 days)
  Heart rate will be continuously assessed during exercise
Systolic and diastolic blood pressure during exercise (mmHg) | Acute/chronic effects (0 and 7 days)
  Blood pressure will be assessed during high intensity intervals.
Plasma glucose concentrations (mg dL-1) | Acute/chronic effects (0 and 7 days)
  Serum concentrations of glycemia (in mg per dL) after 8-hour fasting
Plasma insulin concentrations (µIU mL-1) | Acute/chronic effects (0 and 7 days)
  Serum concentrations of insulin after 8-hour fasting

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR